CLINICAL TRIAL: NCT07112586
Title: Evaluation of Intradermal Exosome Injection in Treatment of Male Androgenetic Alopecia: A Clinical and Immunohistochemical Study
Brief Title: Evaluation of Exosomes Injection in Treatment of Male Androgenetic Alopecia: Clinical and Immunohistochemical Study
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fmasu MD 12 20242025
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Males 18-40 years old with androgenetic alopecia (Experimental): Males with androgenetic alopecia willing to do mesotherapy sessions
  Interventions: Drug: Plasma derived exosomes

INTERVENTIONS:
Drug: Plasma derived exosomes — Exosomes derived from patients' plasma, centrifuged at high speeds multiple times

SUMMARY:
Intradermal injection of exosomes in treatment of male androgenetic alopecia, clinically and using a immunohistochemical marker

ELIGIBILITY:
Inclusion Criteria:

- Androgenetic Alopecia Grades 1-4

Exclusion Criteria:

* blood diseases Receiving other treatments History of malignancy or allergic reaction to exosomes

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 15 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Terminal to vellus hair ratio improvement | One year
  Counting the terminal and vellus hair counts and calculating the ratio, and comparing it between different study sessions and at follow-ups

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Univeristy Faculty of medicine, Cairo, Abbasia, Egypt